CLINICAL TRIAL: NCT06222814
Title: Evaluation of the Results of Two Different Methods in Management of Antero-lateral Instability of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Abdelkareem, Assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-23-12-12MS
Record Dates: First submitted 2024-01-01; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reconstruction group (Active Comparator): Patients with ACL injury and antero-lateral knee instability undergo ACL reconstruction combined with anterolateral ligament reconstruction using peroneus longus autograft
  Interventions: Procedure: ACL reconstruction combined with anterolateral ligament reconstruction using peroneus longus autograft
- Tenodesis group (Active Comparator): Patients with ACL injury and antero-lateral knee instability undergo ACL reconstruction combined with extra-articular tenodesis (Modified Lemaire).
  Interventions: Procedure: ACL reconstruction combined with extra-articular tenodesis (Modified Lemaire)

INTERVENTIONS:
Procedure: ACL reconstruction combined with anterolateral ligament reconstruction using peroneus longus autograft — ACL reconstruction combined with anterolateral ligament reconstruction using peroneus longus autograft
  Arms: Reconstruction group
Procedure: ACL reconstruction combined with extra-articular tenodesis (Modified Lemaire) — ACL reconstruction combined with extra-articular tenodesis (Modified Lemaire)
  Arms: Tenodesis group

SUMMARY:
This randomized clinical study will be conducted to compare the results of anterior cruciate ligament reconstruction (ACLR) combined with either anterolateral ligament reconstruction using peroneus longus autograft or extra-articular tenodesis (Modified Lemaire) in management of antero-lateral instability of the knee

DETAILED DESCRIPTION:
Patients will undergo an anatomic ACLR in a standardized fashion by the same team of surgeons. They are randomly divided into 2 groups either ACLR plus ALL reconstruction or ACLR combined with LET in a 1:1 ratio. There are multiple graft options for ACL-R, but here for the study, the hamstring autograft is harvested following the traditional technique. The graft is measured and bony tunnels are drilled. An anatomical reconstruction technique is used in all cases.

In group A: the surgeon will harvest peroneus longus graft, then sutured to the double bundle hamstring graft. The graft diameters are measured and recorded. The graft is pulled through the femoral tunnel and passed through the tibial tunnel. The single portion of the graft is passed freely through the tibial and femoral tunnels until the quintuple graft portion occupies both tunnels. The graft is then pulled, and an interference screw (Smith & Nephew Endoscopy) is fixed to the femur. The next step is to fix the inferior end of the quintuple graft to the tibia after pre-tensioning. After tibial fixation, the remaining PL is passed through the subcutaneous and ALL tunnels. The ligament is fixed under traction, mild valgus stress, and 30' of flexion 1.5 cm from the joint line into a midpoint between Gerdy's tubercle and the fibular head.

In group B: the surgeon will use a triple STG hamstring (6- strands) tendon graft. The graft diameters are measured and recorded.

Then, LET is performed in a standardized fashion as described in the modified Lemaire technique. LET is fixed with interference screws (Smith & Nephew Endoscopy). Femoral and tibial fixations are performed with bio-absorbable interference screws (Smith & Nephew Endoscopy).

ELIGIBILITY:
Inclusion Criteria:

1. The ACL deficient knee was clinically manifested by physical examination and confirmed by MRI.
2. Age 18-45 years, skeletally mature patient.
3. A positive pivot shift test of at least grade II is required (significant anterolateral instability).

Exclusion Criteria:

1. Multiple ligament injuries or a polytraumatized patient
2. Revision cases.
3. Generalized laxity.
4. Symptomatic articular cartilage defect requiring treatment; Outerbridge > grade II.
5. More than three degrees of varus or valgus malalignment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Functional results of knee stability and return to normal activity | 12 months postoperatively
  IKDC (International Knee Documentation Committee) subjective knee evaluation form

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman Hafez, MD, Study Chair — Professor
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Azab H, Abdelkareem O, Hafez AR, Elsayed M, Ali M. Comparative study between lateral extra-articular tenodesis versus anterolateral ligament reconstruction in combination with anterior cruciate ligament reconstruction. J Orthop Surg Res. 2026 Jan 17. doi: 10.1186/s13018-025-06561-x. Online ahead of print. PMID 41547885